CLINICAL TRIAL: NCT05421091
Title: Special Drug Use-results Surveillance of Scemblix Tablets (Resistant or Intolerant Chronic Myeloid Leukemia , CABL001A1401)
Brief Title: Special Drug Use-results Surveillance of Scemblix Tablets
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CABL001A1401
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Chronic Myeloid Leukemia
Keywords: chronic myeloid leukemia; CML; Scemblix Tablets; Asciminib; resistant or intolerant CML
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — asciminib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Asciminib: Patients prescribed with Asciminib
  Interventions: Other: Asciminib

INTERVENTIONS:
Other: Asciminib — Prospective observational study. There is no treatment allocation. Patients prescribed with asciminib are eligible to enroll into this study.

SUMMARY:
Uncontrolled, central registration system, all-case, multicenter, special drug use-results surveillance.

DETAILED DESCRIPTION:
The objective of this study is to collect data on the occurrence, severity, clinical courses of the safety specifications of asciminib, identify factors etc. involved in occurrence and assess its clinical safety inresistant/intolerant chronic myelogenous leukemia patients during an observational period of 48 weeks from the start of treatment with asciminib.

ELIGIBILITY:
Inclusion Criteria:

* patients treated with asciminib in Japan.

Exclusion Criteria:

NA

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with asciminib
Sampling Method: Non-Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Type, frequency, seriousness and severity of adverse event (AE)/treatment-related AE of the safety specifications | Up to 48 Weeks
  For the safety specifications (myelosuppression, infections, QT interval prolongation, pancreatitis, vascular occlusive events, photosensitivity), type, frequency AE, seriousness, severity of adverse event (AE)/treatment-related AE will be collected
AEs leading to interruption/discontinuation of the safety specifications | Up to 48 Weeks
  For the safety specifications (myelosuppression, infections, QT interval prolongation, pancreatitis, vascular occlusive events, photosensitivity), AEs leading to interruption/discontinuation will be collected
Number of patients with changes in relevant laboratory parameters for the safety specifications | Up to 48 Weeks
  For the safety specifications (myelosuppression, infections, QT interval prolongation, pancreatitis, vascular occlusive events, photosensitivity), number of patients with changes in relevant laboratory parameters will be collected
Frequency of AEs/Treatment-related AEs by patient characteristic factor | Up to 48 Weeks
  Frequency of AEs/Treatment-related AEs by patient characteristic factor will be collected

SECONDARY OUTCOMES:
Type, frequency, seriousness, severity of AEs/treatment-related AEs of the safety analysis set | Up to 48 Weeks
  Type, frequency, seriousness, severity of AEs/treatment-related AEs of the safety analysis set will be collected
AEs leading to interruption/discontinuation in the safety analysis set | Up to 48 Weeks
  AEs leading to interruption/discontinuation in the safety analysis set will be collected
Frequency of AEs/treatment-related AEs summarized by patient characteristic factor | Up to 48 Weeks
  Frequency of AEs/treatment-related AEs summarized by patient characteristic factor will be collected
Type, frequency, seriousness, severity of AEs/treatment-related AEs in patients with special characteristics | Up to 48 Weeks
  Type, frequency, seriousness, severity of AEs/treatment-related AEs in patients with special characteristics (patients with concurrent renal impairment/hepatic impairment/cardiac impairment, elderly, children, pregnant/parturient women) will be collected
AEs leading to interruption/discontinuation in patients with special characteristics | Up to 48 Weeks
  AEs leading to interruption/discontinuation in patients with special characteristics (patients with concurrent renal impairment/hepatic impairment/cardiac impairment, elderly, children, pregnant/parturient women) will be collected
Type, frequency, seriousness, severity and outcome of AEs/treatment-related AEs by treatment line | Up to 48 Weeks
  Type, frequency, seriousness, severity and outcome of AEs/treatment-related AEs by treatment line will be collected
Factors affecting occurrence of AEs by treatment line | Up to 48 Weeks
  Factors affecting occurrence of AEs by treatment line will be collected
AEs leading to interruption/discontinuation by treatment line | Up to 48 Weeks
  AEs leading to interruption/discontinuation by treatment line will be collected
Major molecular response (MMR) rates | Week 12, Week 24, Week 48
  Major molecular response is defined as BCR-ABL1 International Scale value ≤ 0.1%.
  BCR-ABL1: translocation-produced fusion gene
MMR rates by Week 48 by patient characteristics factor | Up to 48 Weeks
  Major molecular response (MMR) is defined as BCR-ABL1 International Scale value ≤ 0.1%.
  BCR-ABL1: translocation-produced fusion gene
MR4.0 and MR4.5 rates | Week 12, Week 24 and Week 48
  MR4.0 and MR4.5 rates are defined as :
  * MR4.0: BCR-ABL1 International Scale value ≤ 0.01%
  * MR4.5: BCR-ABL1 International Scale value ≤ 0.0032%
  BCR-ABL1: translocation-produced fusion gene
Complete cytogenetic response (CCyR) rates | Week 12, Week 24 and Week 48
  This study will collect complete cytogenetic response (CCyR), which is defined as a state of Ph+ metaphase cell disappearance, i.e. Ph+ cell = 0%.
Complete hematological response (CHR) rates | Week 12, Week 24 and Week 48
  This study will collect complete hematological response (CHR), which is defined as meeting the following 6 criteria.
  1. White blood cell count < 10,000/µL
  2. Platelet count < 450,000/µL
  3. No blast cell and promyelocyte in peripheral blood
  4. Myelocyte + metamyelocyte in peripheral blood = 0%
  5. Basophil < 5%
  6. No spleen and liver swelling, and no extramedullary lesion
Rate of patients with BCR-ABL1 gene mutations | Up to 48 Weeks
  This study will collect the rate of patients with BCR-ABL1 gene mutations
MMR rates by Week 48 in patients with special characteristics | Week 48
  This study will collect major molecular response (MMR) rates by Week 48 in patients with special characteristics (patients with concurrent renal impairment/hepatic impairment/cardiac impairment, elderly, children, pregnant/parturient women)
MMR rates by treatment line | Week 12, Week 24 and Week 48
  This study will collect major molecular response (MMR) rates by treatment line
MR4.0 and MR4.5 rates by treatment line | Week 12, Week 24 and Week 48
  MR4.0 and MR4.5 rates are defined as :
  * MR4.0: BCR-ABL1 International Scale value ≤ 0.01%
  * MR4.5: BCR-ABL1 International Scale value ≤ 0.0032%
  BCR-ABL1: translocation-produced fusion gene
CCyR rates by treatment line | Week 12, Week 24 and Week 48
  This study will collect complete cytogenetic response (CCyR), which is defined as a state of Ph+ metaphase cell disappearance, i.e. Ph+ cell = 0%.
CHR rates by treatment line | Week 12, Week 24 and Week 48
  This study will collect complete hematological response (CHR), which is defined as meeting the following 6 criteria.
  1. White blood cell count < 10,000/µL
  2. Platelet count < 450,000/µL
  3. No blast cell and promyelocyte in peripheral blood
  4. Myelocyte + metamyelocyte in peripheral blood = 0%
  5. Basophil < 5%
  6. No spleen and liver swelling, and no extramedullary lesion

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (192):
- Japan (192):
  - Novartis Investigative Site, Anjo, Aichi-ken
  - Novartis Investigative Site, Ichinomiya, Aichi-ken
  - Novartis Investigative Site, Kasugai, Aichi-ken
  - Novartis Investigative Site, Komaki, Aichi-ken
  - Novartis Investigative Site, Kōnan, Aichi-ken
  - Novartis Investigative Site, Nagakute, Aichi-ken
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Seto, Aichi-ken
  - Novartis Investigative Site, Toyoake, Aichi-ken
  - Novartis Investigative Site, Toyohashi, Aichi-ken
  - Novartis Investigative Site, Tōkai, Aichi-ken
  - Novartis Investigative Site, Yatomi, Aichi-ken
  - Novartis Investigative Site, Ōdate, Akita
  - Novartis Investigative Site, Funabashi, Chiba
  - Novartis Investigative Site, Ichihara, Chiba
  - Novartis Investigative Site, Ichikawa, Chiba
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Kisarazu, Chiba
  - Novartis Investigative Site, Matsudo, Chiba
  - Novartis Investigative Site, Narita, Chiba
  - Novartis Investigative Site, Matsuyama, Ehime
  - Novartis Investigative Site, Tōon, Ehime
  - Novartis Investigative Site, Yoshida-gun, Fukui
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Kurume, Fukuoka
  - Novartis Investigative Site, Yanagawa, Fukuoka
  - Novartis Investigative Site, Aizu-Wakamatsu, Fukushima
  - Novartis Investigative Site, Fukushima, Fukushima
  - Novartis Investigative Site, Iwaki, Fukushima
  - Novartis Investigative Site, Gifu, Gifu
  - Novartis Investigative Site, Sekimachi, Gifu
  - Novartis Investigative Site, Takayama, Gifu
  - Novartis Investigative Site, Fujioka, Gunma
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Ōta, Gunma
  - Novartis Investigative Site, Fukuyama, Hiroshima
  - Novartis Investigative Site, Mihara, Hiroshima
  - Novartis Investigative Site, Asahikawa, Hokkaido
  - Novartis Investigative Site, Hakodate, Hokkaido
  - Novartis Investigative Site, Iwamizawa, Hokkaido
  - Novartis Investigative Site, Kushiro, Hokkaido
  - Novartis Investigative Site, Obihiro, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Akashi, Hyōgo
  - Novartis Investigative Site, Amagasaki, Hyōgo
  - Novartis Investigative Site, Himeji, Hyōgo
  - Novartis Investigative Site, Kakogawa-shi, Hyōgo
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Nishinomiya, Hyōgo
  - Novartis Investigative Site, Sumoto, Hyōgo
  - Novartis Investigative Site, Toyooka, Hyōgo
  - Novartis Investigative Site, Higashiibaraki-gun, Ibaraki
  - Novartis Investigative Site, Hitachi, Ibaraki
  - Novartis Investigative Site, Ishioka, Ibaraki
  - Novartis Investigative Site, Koga, Ibaraki
  - Novartis Investigative Site, Tsuchiura, Ibaraki
  - Novartis Investigative Site, Tsukuba, Ibaraki
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Nanao, Ishikawa-ken
  - Novartis Investigative Site, Nomi, Ishikawa-ken
  - Novartis Investigative Site, Kitakami, Iwate
  - Novartis Investigative Site, Morioka, Iwate
  - Novartis Investigative Site, Shiwa-gun, Iwate
  - Novartis Investigative Site, Kita-gun, Kagawa-ken
  - Novartis Investigative Site, Takamatsu, Kagawa-ken
  - Novartis Investigative Site, Kanoya, Kagoshima-ken
  - Novartis Investigative Site, Kirishima, Kagoshima-ken
  - Novartis Investigative Site, Kamakura, Kanagawa
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Yamato, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kochi, Kochi
  - Novartis Investigative Site, Kumamoto, Kumamoto
  - Novartis Investigative Site, Fukuchiyama, Kyoto
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Maizuru, Kyoto
  - Novartis Investigative Site, Tsu, Mie-ken
  - Novartis Investigative Site, Yokkaichi, Mie-ken
  - Novartis Investigative Site, Ishinomaki, Miyagi
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Miyakonojō, Miyazaki
  - Novartis Investigative Site, Nobeoka, Miyazaki
  - Novartis Investigative Site, Nagano, Nagano
  - Novartis Investigative Site, Saku, Nagano
  - Novartis Investigative Site, Suwa, Nagano
  - Novartis Investigative Site, Isahaya, Nagasaki
  - Novartis Investigative Site, Nagasaki, Nagasaki
  - Novartis Investigative Site, Ikoma, Nara
  - Novartis Investigative Site, Kashihara, Nara
  - Novartis Investigative Site, Tenri, Nara
  - Novartis Investigative Site, Jōetsu, Niigata
  - Novartis Investigative Site, Minamiuonuma, Niigata
  - Novartis Investigative Site, Nagaoka, Niigata
  - Novartis Investigative Site, Shibata, Niigata
  - Novartis Investigative Site, Yufu, Oita Prefecture
  - Novartis Investigative Site, Kurashiki, Okayama-ken
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Tsuyama, Okayama-ken
  - Novartis Investigative Site, Nago, Okinawa
  - Novartis Investigative Site, Naha, Okinawa
  - Novartis Investigative Site, Shimajiri-Gun, Okinawa
  - Novartis Investigative Site, Hirakata, Osaka
  - Novartis Investigative Site, Izumisano, Osaka
  - Novartis Investigative Site, Kawachi-Nagano, Osaka
  - Novartis Investigative Site, Moriguchi, Osaka
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Ōsaka-sayama, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Takatsuki, Osaka
  - Novartis Investigative Site, Tondabayashi, Osaka
  - Novartis Investigative Site, Toyonaka, Osaka
  - Novartis Investigative Site, Karatsu, Saga-ken
  - Novartis Investigative Site, Saga, Saga-ken
  - Novartis Investigative Site, Asaka, Saitama
  - Novartis Investigative Site, Fukaya, Saitama
  - Novartis Investigative Site, Hidaka, Saitama
  - Novartis Investigative Site, Iruma-gun, Saitama
  - Novartis Investigative Site, Kawagoe, Saitama
  - Novartis Investigative Site, Koshigaya, Saitama
  - Novartis Investigative Site, Sayama, Saitama
  - Novartis Investigative Site, Tokorozawa, Saitama
  - Novartis Investigative Site, Kusatsu, Shiga
  - Novartis Investigative Site, Moriyama, Shiga
  - Novartis Investigative Site, Nagahama, Shiga
  - Novartis Investigative Site, Ōmihachiman, Shiga
  - Novartis Investigative Site, Izumo, Shimane
  - Novartis Investigative Site, Masuda, Shimane
  - Novartis Investigative Site, Matsue, Shimane
  - Novartis Investigative Site, Hamamatsu, Shizuoka
  - Novartis Investigative Site, Iwata, Shizuoka
  - Novartis Investigative Site, Izunokuni, Shizuoka
  - Novartis Investigative Site, Shimada, Shizuoka
  - Novartis Investigative Site, Shizuoka, Shizuoka
  - Novartis Investigative Site, Sunto Gun, Shizuoka
  - Novartis Investigative Site, Sano, Tochigi
  - Novartis Investigative Site, Shimotsuke, Tochigi
  - Novartis Investigative Site, Komatsushimachō, Tokushima
  - Novartis Investigative Site, Okuno, Tokushima
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Chiyoda-ku, Tokyo
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Itabashi Ku, Tokyo
  - Novartis Investigative Site, Komae, Tokyo
  - Novartis Investigative Site, Koto Ku, Tokyo
  - Novartis Investigative Site, Meguro City, Tokyo
  - Novartis Investigative Site, Meguro-ku, Tokyo
  - Novartis Investigative Site, Minato Ku, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Mitaka, Tokyo
  - Novartis Investigative Site, Musashino, Tokyo
  - Novartis Investigative Site, Nerima-ku, Tokyo
  - Novartis Investigative Site, Ōme, Tokyo
  - Novartis Investigative Site, Shibuya City, Tokyo
  - Novartis Investigative Site, Shinagawa Ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Suginami, Tokyo
  - Novartis Investigative Site, Sumida-ku, Tokyo
  - Novartis Investigative Site, Tachikawa, Tokyo
  - Novartis Investigative Site, Yonago, Tottori
  - Novartis Investigative Site, Tonami, Toyama
  - Novartis Investigative Site, Toyama, Toyama
  - Novartis Investigative Site, Kinokawa, Wakayama
  - Novartis Investigative Site, Sakata, Yamagata
  - Novartis Investigative Site, Ube, Yamaguchi
  - Novartis Investigative Site, Chūō, Yamanashi
  - Novartis Investigative Site, Kofu, Yamanashi
  - Novartis Investigative Site, Akita
  - Novartis Investigative Site, Aomori
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Fukui
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Fukushima
  - Novartis Investigative Site, Gifu
  - Novartis Investigative Site, Hiroshima
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Miyazaki
  - Novartis Investigative Site, Nagasaki
  - Novartis Investigative Site, Nara
  - Novartis Investigative Site, Niigata
  - Novartis Investigative Site, Okayama
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Ōita
  - Novartis Investigative Site, Saitama
  - Novartis Investigative Site, Tochigi
  - Novartis Investigative Site, Tokushima
  - Novartis Investigative Site, Toyama
  - Novartis Investigative Site, Wakayama
  - Novartis Investigative Site, Yamagata

IPD SHARING:
Plan to Share IPD: No